CLINICAL TRIAL: NCT01649245
Title: Efficacy and Safety of a Hansenula-derived Pegylated Interferon α2a (Reiferon Retard®) in Treatment of Patients With Chronic Hepatitis C Virus Infection: A National Multi-center Phase IV Open Label Non-Randomized Trial
Brief Title: Hansenula-derived Pegylated Interferon in Treatment of Patients With Chronic Hepatitis C
Acronym: HAPIC
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: MinaPharm Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HAPIC Trial
Record Dates: First submitted 2012-07-20; First posted 2012-07-25 (Estimated); Last update posted 2013-01-15 (Estimated); Status verified 2013-01

CONDITIONS: Chronic Hepatitis C
Keywords: Chronic hepatitis C; Egyptian patients; pegylated interferon; Ribavirin; Reiferon retard
MeSH Terms: conditions — Hepatitis C, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Reiferon retard plus ribavirin (Experimental): Eligible subjects will be treated with Reiferon Retard® 160 µg weekly by subcutaneous injection for 48 weeks, together with weight-based oral ribavirin (1200 mg/day if body weight is >75 kg and 1000 mg/day if body weight is ≤ 75 kg) in divided doses
  Interventions: Drug: Reiferon retard

INTERVENTIONS:
Drug: Reiferon retard — Eligible subjects will be treated with Reiferon Retard® 160 µg weekly by subcutaneous injection for 48 weeks, together with weight-based oral ribavirin (1200 mg/day if body weight is >75 kg and 1000 mg/day if body weight is ≤ 75 kg) in divided doses.
  Other Names: Pegylated interferon α 2a

SUMMARY:
It is a multi-center study of the efficacy of a new Pegylated Hansenula-derived recombinant interferon α 2a (Reiferon Retard® 160 µg once weekly in combination with ribavirin in treatment of Egyptian patients with chronic hepatitis C for 48 weeks.

hepatitis C virus (HCV) viral load will be assessed during therapy at weeks 12, 24 and end of treatment, as well as 24 weeks after therapy is completed.

DETAILED DESCRIPTION:
Multicenter , Phase IV, open labeled, non-randomized trial to assess the Efficacy of Hansenula-derived recombinant pegylated interferon α 2a (Reiferon Retard® in treatment of naïve chronic hepatitis c virus Egyptian patients.

Each participant will be subject to thorough history taking, complete clinical examination, Biochemical laboratory and hematological tests, U/S imaging as well as histologic assessment of liver disease stage and severity to ensure his/her eligibility to be enrolled in the study according to predetermined inclusion and exclusion criteria .

Eligible subjects will be treated with Reiferon Retard® 160 µg once weekly by subcutaneous injection for 48 weeks treatment plus weight-based Ribavirin orally (1200 mg/kg daily for those > 75 Kg or 1000mg/Kg daily for those ≤ 75 kg in divided doses). HCV RNA will be assessed at week 12 of initiation of therapy to identify Early Virologic Response (EVR), at week 24 to identify breakthrough viremia, at week 48 to identify End of treatment Response (ETR), and at week 72 to identify Sustained Virologic Response (SVR).

All subjects will be followed up during the study as described in the table below (Section 4 Study Design).

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18 and < 60.
2. BMI ≤ 30
3. Liver biopsy showing chronic hepatitis with significant fibrosis (F2 and F3 using Metavir scoring system) regardless of aminotransferase elevations.
4. F1 stage (by Metavir scoring system) with elevated aminotransferases.
5. Compensated liver disease; serum bilirubin < 1.5 mg/dl, INR no more than 1.5, serum albumin ≥ 3.5 g/dl, platelet count ≥ 1000 cmm, and no evidence of hepatic decompensation (hepatic encephalopathy or ascites).
6. Acceptable hematological and biochemical indices (hemoglobin ≥ 11g/dl; total leukocytic count ≥ 3000/cmm, absolute neutrophil count ≥ 1500/cmm and serum creatinine < 1.97 mg/dl.
7. Willing to be treated and to adhere to treatment requirements.

Exclusion Criteria:

1. Major uncontrolled depressive illness.
2. Solid organ transplantation.
3. Autoimmune conditions, known to be exacerbated by peginterferon and ribavirin.
4. Untreated thyroid disease.
5. Pregnant or unwilling to comply with adequate contraception.
6. Severe concurrent medical disease, such as severe hypertension, heart failure, significant coronary artery disease, poorly controlled diabetes (HbA1C > 8.5 %), and chronic obstructive pulmonary disease.
7. Known hypersensitivity to drugs used to treat HCV.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 5000 (Estimated)
Dates: Start 2012-08; Primary Completion 2014-08 (Estimated); Study Completion 2014-08 (Estimated)

PRIMARY OUTCOMES:
Sustained Virologic Response (SVR) | Assessed 24 weeks after the end of treatment
  Sustained Virologic Response (SVR) is assessed by measurement of HCV RNA viral load 24 weeks after the end of Therapy.
  SVR is defined as undetectable HCV RNA 24 weeks after the end of therapy.

SECONDARY OUTCOMES:
Complete Early Virologic Response (cEVR) | At week 12 of therapy
  Complete Early Virologic Response (cEVR)is defined as undetectable HCV RNA at week 12 of therapy.
End of Treatment Response (ETR) | at the end of therapy (48 weeks from initiation of therapy
  ETR is defined as undetectable HCV RNA at the end of therapy (at week 48)
Safety | Throughout the duration of therapy (48weeks)
  Drug safety will be monitored throughout the treatment duration (48 weeks), and any moderate to severe adverse events will be reported

CONTACTS AND LOCATIONS:
Overall Officials: Imam Waked, MD, Principal Investigator — National Liver Institute, Egypt; Gamal Esmat, MD, Principal Investigator — Faculty of Medicine - Cairo University - Egypt; Hassan Hamdy, MD, Principal Investigator — Faculty of Medicine - Ain Shams University - Egypt; Mohamed kohla, MD, Study Director — National Liver Institute, Egypt
Locations (1):
- National Liver Institute, Shebin El-Kom, Monufia Governorate, Egypt